CLINICAL TRIAL: NCT03718975
Title: Quality Control of CE-Certified Phonak Hearing Aids - 2018_28
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Sonova2018_28
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Hearing Loss; Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Successor of Phonak Audéo B90 (Experimental): The successor of the Phonak Audéo B90 is a Receiver-in-the-canal Hearing aid with direct connectivity functionality from Phonak which will be fitted to the participants individual Hearing loss.
  Interventions: Device: Successor of Phonak Audéo B90
- Phonak Audéo B90 (Active Comparator): The Phonak Audéo B90 is the most recent Receiver-in-the-canal Hearing aid from Phonak which will be fitted to the participants individual Hearing loss.
  Interventions: Device: Phonak Audéo B90

INTERVENTIONS:
Device: Successor of Phonak Audéo B90 — Successor of the most recent Receiver in the canal (RIC) Hearing aid form Phonak which will be fitted to the participants individual Hearing loss.
  Arms: Successor of Phonak Audéo B90
Device: Phonak Audéo B90 — The Phonak Audéo B90 is the most recent Receiver-in-the-canal Hearing aid from Phonak which will be fitted to the participants individual Hearing loss.
  Arms: Phonak Audéo B90

SUMMARY:
Phonak Hearing Systems pass through different development and study stages. At an early stage, feasibility studies are conducted to investigate new algorithms, features and functions in an isolated manner. If the benefit is proven, their performance is then investigated regarding interdependency between all available algorithms, features and functions running in parallel in a hearing aid (pivotal/pre-validation studies) and, as a result, they get optimized. Afterwards, and prior to product launch, the Phonak Hearing Systems undergo a final quality control in terms of clinical trials. This is a pre-validation study, investigating optimized algorithms, features, functions and wearing comfort. This will be a clinical investigation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

DETAILED DESCRIPTION:
In this study a comparison with two CE-labeled Phonak Receiver-in-the-canal (RIC) devices is done. The experimental device and the active comparator will be compared regarding Sound Quality perception and speech intelligibility in Quiet and in Noise. The experimental device contains direct connectivity functionality which will be investigated in terms of streamed Audio quality, streaming stability and Usability preferences of functions and Features which are related to direct connectivity. The active comparator device does not contain direct streaming functionality. This will be a clinical investigation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* Adult hearing impaired persons (minimum age: 18 years, mild to moderate Hearing loss) without hearing aid experience
* Good written and spoken (Swiss) German language skills
* Healthy outer ear
* Ability to fill in a questionnaire (p/eCRF) conscientiously
* willingness to wear Receiver in the canal hearing aids
* Informed Consent as documented by signature
* owning a compatible smartphone

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments in Stäfa (Switzerland)
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Known psychological problems
* Central hearing disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-12-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of subjective acceptance of the default Hearing aid setting | 10 weeks
  The Primary Outcome measure of this study is the comparison of the default Hearing aid Fitting (first fit) in regard of the subjective acceptance rating between the experimental device and the active comparator (non-inferiority test design). The first fit acceptance will be measured via subjective satisfaction rating of different dimensions concerning sound quality perception and loudness perception (Scale of satisfaction rating ranging from 0% to 100%).

SECONDARY OUTCOMES:
Subjective Sound Quality rating of streamed telephone call (experimental device only) | 10 weeks
  The secondary Outcome measure of this study is the Evaluation of the perceived Sound Quality (rated via subjective satisfaction rating) of the streamed telephone signal, which will be streamed between a smartphone and the experimental device.

OTHER OUTCOMES:
Evaluation of Speech intelligibility in noise | 10 weeks
  Another Outcome measure of this study is the Evaluation of speech understanding in noise of the experimental device and the active comparator. Speech understanding in noise will be evaluated with an objective and validated test procedure, the Outcome measure will be the Signal-to-noise ration (SNR) in dB.
Evaluation of Speech intelligibility in quiet | 10 weeks
  Another Outcome measure of this study is the Evaluation of speech understanding in quiet of the experimental device and the active comparator. Speech understanding in quiet will be evaluated with an objective and validated test procedure, the Outcome measure will be the speech intelligibility in % at certain Levels of loudness.
Evaluation of the Bluetooth stability (experimental device only) | 10 weeks
  Another outcome measure of this study is the investigation of bluetooth stability of the experimental device in terms of connection losses and interruptions. The bluetooth stability will be measured via interview and questionnaires during and after a home trial for the experimental device only. The active comparator device does not have Bluetooth Technology.
Evaluation of Usability preferences (experimental device only) | 10 weeks
  Another Outcome measure is the qualitative rating of user preferences when using direct connectivity Technology in Terms of streaming an audio signal from an external device with Bluetooth Technology to the experimental device. The user preferences will investigated via rating scales client on a questionnaire during a home trial period

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No